CLINICAL TRIAL: NCT04947813
Title: Association Analysis Between Variants of COL4A3/COL4A4/COL4A5 and Alport Syndrome in the Han Chinese Population
Brief Title: Genotype-Phenotype Correlations in Patients With Alport Syndrome
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2020-102-1
Record Dates: First submitted 2021-06-03; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-05

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alport syndrome (AS) is caused by pathogenic variants in the type IV collagen genes COL4A3, COL4A4, and COL4A5. This study aims to enroll families and patients with a history of renal hematuria in 27 hospitals and detect these three genes for AS screening. This study also aims to analysis the effect of COL4A3/COL4A4/COL4A5 genotype on the development of kidney disease.

DETAILED DESCRIPTION:
Alport syndrome (AS) is a genetically and phenotypically heterogeneous disorder caused by the mutations in the type IV collagen genes COL4A3, COL4A4, and COL4A5. In this study, next generation sequencing is used to screen AS on 8165 participants enrolled from families and patients with a history of renal hematuria in 27 hospitals of China Huadong Region. Genotype (variants in COL4A3/COL4A4/COL4A5)-phenotype (onset age of hearing loss, nephroticrange proteinuria, decline of eGFR, kidney survival and onset age of CKD5) correlations in AS were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: up to 99 Years (Child, Adult, Older Adult)
2. Sex: All;
3. Families and patients with a history of renal hematuria;
4. Those who signed the informed consent.

Exclusion Criteria:

1. Polycystic kidney disease, hypertensive nephropathy, etc.;
2. Kidney biopsy is diagnosed as other primary/secondary kidney disease without type IV collagen-related kidney disease, including IgA nephropathy, membranous nephropathy, lupus nephritis, etc.
3. Incomplete medical history or clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Xinhua Hospital, Shanghai Jiao Tong University School of Medicine and other 26 hospitals of China Huadong Region.
Sampling Method: Non-Probability Sample
Enrollment: 8165 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification COL4A3/COL4A4/COL4A5 variants of Alport Syndrome | Up to 240 weeks
  To characterize the variants of COL4A3/COL4A4/COL4A5 in patients with Alport syndrome over the course of up to 240 weeks

SECONDARY OUTCOMES:
Identification genotype-phenotype correlations of Alport Syndrome | Up to 240 weeks
  Exploring correlations between variants of COL4A3/COL4A4/COL4A5 and the clinical robustness including onset age of hearing loss, nephroticrange proteinuria, decline of eGFR, kidney survival and onset age of CKD5 in Alport syndrome patients

CONTACTS AND LOCATIONS:
Locations (1):
- China Xinhua Hospital, Shanghai Jiao Tong University School of Medicine., Shanghai, China